CLINICAL TRIAL: NCT05813288
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Dexpramipexole Administered Orally for 52 Weeks in Participants With Severe Eosinophilic Asthma
Brief Title: A Study to Assess the Effect of Dexpramipexole in Adolescents and Adults With Severe Eosinophilic Asthma (EXHALE-3)
Acronym: EXHALE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program stopped due to the benefit risk profile no longer supports further development in the intended patient population.
Sponsor: Areteia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-DEX-22-02; 2023-503693-20 (EudraCT Number)
Record Dates: First submitted 2023-03-27; First posted 2023-04-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Asthma; Asthma; Eosinophilic; Asthma
Keywords: Exacerbations; Severe Asthma; Dexpramipexole; EXHALE; Areteia; EXHALE-3; Uncontrolled Asthma; Asthma Attack
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg BID (Experimental): Dexpramipexole 150 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- 75 mg BID (Experimental): Dexpramipexole 75 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- Placebo (Placebo Comparator): Placebo oral tablet taken twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpramipexole Dihydrochloride — Oral administration of dexpramipexole tablet
  Arms: 150 mg BID; 75 mg BID
Drug: Placebo — Oral administration of placebo tablet
  Arms: Placebo

SUMMARY:
The objective of this clinical study is to investigate the safety, tolerability, and efficacy of dexpramipexole in participants with inadequately controlled severe eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and assent form, as appropriate.
2. Male or female ≥12 years of age at Screening Visit 1.

   Asthma-related criteria
3. Documented physician diagnosis of asthma for ≥12 months prior to Screening Visit 1.
4. Eosinophil count of ≥0.30x10⁹/L at Screening Visit 1. If the initial value is between 0.250x10⁹/L to 0.299x10⁹/L, then this may be repeated once at an unscheduled visit (prior to Screening Visit 2).
5. Treatment of asthma, participants must satisfy all the below (items a to c):

   1. Participants who have received asthma controller medication with medium or high dose inhaled corticosteroids (ICS ≥500 μg/day fluticasone propionate dry powder formulation daily or clinically comparable, per GINA 2021) on a regular basis for at least 12 months prior to Screening Visit 1.
   2. Documented treatment with a stable dose of either medium or high dose ICS for at least 3 months prior to Visit 1. The ICS may be contained within an ICS/long-acting β2 agonist (LABA) combination product. Daily oral corticosteroids are an allowed concomitant medication; participants on daily oral corticosteroids must be on a stable dose for 3 months before Screening Visit 1.
   3. Use of one of more additional daily maintenance asthma controller medications according to standard practice of care is required. Use of a stable dose of any additional asthma controller medications must be documented for at least 3 months prior to Screening Visit 1.
6. Pre-BD FEV₁ ≥40% and <80% (<90% for participants 12 to 17 years of age) of predicted at Screening Visit 2.
7. Variable airflow obstruction documented with at least one of the following criteria:

   1. Bronchodilator reversibility at Screening Visit 2, as evidenced by ≥12% and ≥200 mL improvement in FEV₁, 15 to 30 minutes following inhalation of 400 µg (four puffs) of albuterol/salbutamol (≥12% and ≥160 mL for ages 12 to 17). Participants who do not meet the bronchodilator reversibility inclusion criterion but have ≥10% and ≥160 mL reversibility, may repeat the reversibility spirometry assessment once during the Screening period, at an unscheduled visit at least 7 days prior to baseline.
   2. Bronchodilator reversibility, using the criteria above, documented in the past 24 months prior to Screening Visit 1 or during Screening.
   3. Peak flow variation of ≥20% over a 2-week period, documented in the past 24 months prior to Screening Visit 1 or during Screening.
   4. Airflow variability in clinic FEV₁ ≥20% between two consecutive clinic visits, documented in the past 24 months prior to Screening Visit 1.
   5. Airway hyperresponsiveness (provocative concentration causing a 20% fall in FEV₁ of methacholine <8 mg/mL or other clinically relevant bronchoprovocation testing) documented in the past 24 months prior to Screening Visit 1 or during Screening.
8. ACQ-6 ≥1.5 at Screening Visit 2.
9. Documented history of at least two asthma exacerbations requiring treatment with systemic corticosteroids (intramuscular, intravenous, or oral) within the past 12-month period prior to Screening Visit 1.

   General medical history
10. Negative urine pregnancy test for women of childbearing potential (WOCBP; after menarche) at the Screening and Baseline visits.
11. WOCBP must use either of the following methods of birth control, from Screening Visit 1 through the End of Study Visit:

    1. A highly effective form of birth control (confirmed by the investigator). Highly effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective Intrauterine device (IUD), IUD/intrauterine system (IUS), Levonorgestrel Intrauterine system, or oral contraceptive.

       * Or
    2. Two protocol acceptable methods of contraception in tandem.

       Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for ≥12 months prior to the planned date of the Baseline Visit without an alternative medical cause. The following age specific requirements apply:
    3. Women <50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
    4. Women ≥50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

Asthma-related criteria

1. A participant who experiences a severe asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids) at any time from 4 weeks prior to Screening Visit 1.

   Participants who experience an asthma exacerbation during the Screening/Run-in Period may remain in screening and proceed with study visits 14 days after they have completed their course of oral steroids or returned to their pre-Screening Visit maintenance dose of oral steroids and the investigator considers participant has returned to baseline status.
2. Current diagnosis of diseases which may confound interpretation of this study's findings such as allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis, eosinophilic gastrointestinal diseases, hypereosinophilic syndrome, or lung diseases (eg, chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis).
3. Respiratory infection: Upper or lower respiratory tract, sinus, or middle ear infection within the 4 weeks before Screening Visit 1.

   Prohibited medications/procedures
4. Treatment with a biologic investigational drug in the last 5 months prior to Screening Visit 1. Treatment with non-biologic investigational drugs in the previous 30 days or five-half-lives prior to Screening Visit 1, whichever is longer. Treatment with GSK3511294 (long-acting anti-IL-5) in the past 12 months.
5. Treatment with any of the following monoclonal antibody therapies within 120 days prior to Baseline: benralizumab, dupilumab, mepolizumab, reslizumab, omalizumab, tezepelumab, or tralokinumab.
6. Treatment with pramipexole (Mirapex®) within 30 days of Baseline.
7. Treatment with selected drugs known to have a substantial risk of neutropenia in the past 30 days prior to Screening Visit 1.
8. Bronchial thermoplasty procedure in the past 12 months prior to Screening Visit 1 or planned during the coming year.

   General medical history
9. Weight <40 kg at Screening Visit 1.
10. Current smoking within 12 months prior to Screening Visit 1 or a smoking history of >10 pack-years. Smoking includes tobacco, vaping, and/or marijuana use.
11. Known or suspected alcohol or drug abuse
12. Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to Baseline Visit despite anti-hypertensive therapy.
13. History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the 5 years prior to Baseline Visit.
14. History of human immunodeficiency virus (HIV) infection or chronic infection with hepatitis B or C.
15. A helminth parasitic infection diagnosed within 24 weeks prior Screening Visit 1 that has not been treated with or has failed to respond to standard of care (SoC) therapy.
16. Medical or other condition likely to interfere with participant's ability to undergo study procedures, adhere to visit schedule, or comply with study requirements.
17. Known or suspected noncompliance with medication.
18. Unwillingness or inability to follow the procedures outlined in the protocol.

    Clinical safety labs
19. Absolute neutrophil count <2.000x10⁹/L at screening at Screening Visit 1 or Screening Visit 2.
20. Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m² at Screening Visit 2 (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula [Levey et al, 2009] for age ≥18 years at screening; using the Bedside Schwartz [Schwartz and Work, 2009] eGFR formula for age <18).
21. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), >3x the upper limit of normal (ULN), or total bilirubin >2x ULN at Screening Visit 2 confirmed by a repeat abnormal measurement of the relevant value(s), at least 1 week apart.

    Cardiac safety
22. History of New York Heart Association class IV heart failure or last known left ventricular ejection fraction <25%.
23. History of major adverse cardiovascular event (MACE) within 3 months prior to the Baseline Visit.
24. History of cardiac arrhythmia within 3 months prior to Baseline Visit that is not controlled by medication or via ablation.
25. History of long QT syndrome.
26. Corrected QT interval by Fridericia (QTcF) interval >450 ms for males and >470 ms for females at Screening Visit 2 or QTcF ≥480 ms for participants with bundle branch block.
27. Clinically important abnormalities in resting ECG that may interfere with the interpretation of QTcF interval changes at Screening Visit 2, including heart rate <45 beats per minute (bpm) or >100 bpm.

    Pregnancy/Lactation
28. Pregnant women or women breastfeeding.
29. Males who are unwilling to use an acceptable method of birth control during the entire study period (ie, condom with spermicide).
30. Allergy or hypersensitivity to dexpramipexole or any of its components.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Annualized rate of severe asthma exacerbations over 52 weeks. | Day 1 (baseline, pre-dose) through Week 52
  A severe exacerbation was defined as a deterioration of asthma requiring: use of systemic corticosteroids for >=3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids; or death due to asthma.

SECONDARY OUTCOMES:
Absolute Change in pre-bronchodilator forced expiratory volume (Pre-BD FEV₁) from Baseline | Day 1 (baseline, pre-dose), Weeks 36, 44, 52
  The absolute change from baseline in pre-bronchodilator forced expiratory volume, averaged across visits at Weeks 36, 44, and 52.
Mean Change From Baseline at Week 52 in Asthma Control Questionnaire-6 (ACQ-6) (Key Secondary Endpoint) | From randomization to Study Week 52
  Change from baseline in ACQ-6 as compared to placebo at Week 52. The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses
Mean Change From Baseline at Week 52 in Standardized Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ+12) Total Score (Key Secondary Endpoint) | From randomization to Study Week 52
  Mean change from baseline in AQLQ+12 as compared to placebo at Week 52. The AQLQ+12 is a questionnaire that measures the health-related quality of life experienced by asthma subjects. The total score is defined as the average of all 32 questions in the AQLQ+12 questionnaire. AQLQ+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment).
Annualized rate of severe exacerbations requiring an emergency over 52 weeks department visit or hospitalization | Day 1 (baseline, pre-dose), Week 52
Annualized rate of severe exacerbations (AAER) from Week 4 to Week 52. | Week 4 through Week 52
Change in absolute eosinophil count (AEC) | Day 1 (baseline, pre-dose), Weeks 35, 44, and 52
Average change from baseline in forced vital capacity (FVC) | Day 1(baseline, pre-dose), Weeks 36, 44, and 52
FVC, change from baseline at Weeks 4, 12, 20, 28, 36, 44, and 52. | Day 1(baseline, pre-dose), Weeks 4, 12, 20, 28, 36, 44, and 52.
Post-bronchodilator FEV₁, change from baseline to Week 52 | Day 1 (baseline, pre-dose) through Week 52
Time to first severe asthma exacerbation | Up to Week 52
Mean Change From Baseline at Week 52 in Asthma Symptom Diary (ASD) | From randomization to Study Week 52
  The Asthma Symptom Diary comprises of 10 items (5 items in the morning; 5 items in the evening). Asthma symptoms during night time and daytime are recorded by the patient each morning and evening in the daily diary. A daily ASD score is the mean of the 10 items. Responses for all 10 items are required to calculate the daily ASD score; otherwise, it is treated as missing. For the 7-day average asthma symptom score, scoring is done with no imputation using the mean of at least 4 of the 7 daily ASD scores as a mean weekly item score. The 7-day average ASD score ranges from 0 to 4, where 0 indicates no asthma symptoms.
Mean Change From Baseline at Week 52 in EQ-5D-5L | At Study Week 52
  EQ-5D-5L allows subjects to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Wechsler, MD, Principal Investigator — National Jewish Health
Locations (282):
- United States (76):
  - Research Site 30001-287, Mobile, Alabama
  - Research Site 30001-487, Chandler, Arizona
  - Research Site 30001-462, Peoria, Arizona
  - Research Site 30001-322, Surprise, Arizona
  - Research Site 30001-458, Tucson, Arizona
  - Research Site 30001-010, Little Rock, Arkansas
  - Research Site 30001-502, Canoga Park, California
  - Research Site 30001-485, Inglewood, California
  - Research Site 30001-362, Laguna Niguel, California
  - Research Site 30001-497, Los Angeles, California
  - Research Site 30001-500, Northridge, California
  - Research Site 30001-489, Pasadena, California
  - Research Site 30001-501, San Diego, California
  - Research Site 30001-434, San Diego, California
  - Research Site 30001-484, Santa Monica, California
  - Research Site 30001-304, Valencia, California
  - Research Site 30001-305, Valencia, California
  - Research Site 30001-291, Jacksonville, Florida
  - Research Site 30001-318, Maitland, Florida
  - Research Site 30001-311, Miami, Florida
  - Research Site 30001-288, Miami, Florida
  - Research Site 30001-310, Miami, Florida
  - Research Site 30001-329, Miami, Florida
  - Research Site 30001-082, Miami, Florida
  - Research Site 30001-301, Naples, Florida
  - Research Site 30001-348, Ocala, Florida
  - Research Site 30001-331, Orlando, Florida
  - Research Site 30001-293, Orlando, Florida
  - Research Site 30001-312, Pembroke Pines, Florida
  - Research Site 30001-429, Plantation, Florida
  - Research Site 30001-319, Viera, Florida
  - Research Site 30001-452, Dunwoody, Georgia
  - Research Site 30001-483, East Point, Georgia
  - Research Site 30001-366, Lilburn, Georgia
  - Research Site 30001-328, Maywood, Illinois
  - Research Site 30001-535, Westchester, Illinois
  - Research Site 30001-347, Louisville, Kentucky
  - Research Site 30001-437, Alexandria, Louisiana
  - Research Site 30001-286, Lafayette, Louisiana
  - Research Site 30001-313, Marrero, Louisiana
  - Research Site 30001-352, Zachary, Louisiana
  - Research Site 30001-414, Annapolis, Maryland
  - Research Site 30001-472, Farmington Hills, Michigan
  - Research Site 30001-442, Southfield, Michigan
  - Research Site 30001-372, Warren, Michigan
  - Research Site 30001-421, Mankato, Minnesota
  - Research Site 30001-406, Rochester, Minnesota
  - Research Site 30001-522, North Las Vegas, Nevada
  - Research Site 30001-363, Edison, New Jersey
  - Research Site 30001-499, Hamilton, New Jersey
  - Research Site 30001-474, Massena, New York
  - Research Site 30001-455, New York, New York
  - Research Site US-30001-369, New York, New York
  - Research Site 30001-300, Schenectady, New York
  - Research Site 30001-398, Charlotte, North Carolina
  - Research Site 30001-439, Rocky Mount, North Carolina
  - Research Site 30001-413, Cleveland, Ohio
  - Research Site 30001-495, Columbus, Ohio
  - Research Site 30001-327, Philadelphia, Pennsylvania
  - Research Site 30001-414, Franklin, Tennessee
  - Research Site 30001-364, Memphis, Tennessee
  - Research Site 30001-334, Allen, Texas
  - Research Site 30001-090, Austin, Texas
  - Research Site 30001-415, Dallas, Texas
  - Research Site US-30001-418, Frisco, Texas
  - Research Site 30001-299, Houston, Texas
  - Research Site 30001-315, Katy, Texas
  - Research Site 30001-295, McKinney, Texas
  - Research Site 30001-373, Mesquite, Texas
  - Research Site 30001-481, Nederland, Texas
  - Research Site 30001-297, Pearland, Texas
  - Research Site 30001-238, San Antonio, Texas
  - Research Site 30001-377, San Antonio, Texas
  - Research Site 30001-335, Sugar Land, Texas
  - Research Site 30001-333, Pleasant View, Utah
  - Research Site 30001-515, West Valley City, Utah
- Argentina (23):
  - Research Site 30054-035, Buenos Aires
  - Research Site 30054-031, Buenos Aires
  - Research Site 30054-048, Buenos Aires
  - Research Site 30054-045, Buenos Aires
  - Research Site 30054-026, Buenos Aires
  - Research Site 30054-049, Buenos Aires
  - Research Site 30054-050, Buenos Aires
  - Research Site 30054-044, Buenos Aires
  - Research Site 30054-012, Buenos Aires
  - Research Site 30054-021, Buenos Aires
  - Research Site 30054-034, Buenos Aires
  - Research Site 30054-015, Buenos Aires
  - Research Site 30054-024, Buenos Aires
  - Research Site 30054-008, Buenos Aires
  - Research Site -30054-043, Buenos Aires
  - Research Site 30054-054, Concepción del Uruguay
  - Research Site 30054-051, Córdoba
  - Research Site 30054-052, Córdoba
  - Research Site 30054-047, Mendoza
  - Research Site 30054-010, Mendoza
  - Research Site 30054-032, Mendoza
  - Research Site 30054-028, Mendoza
  - Research Site 30054-042, Santa Fe
- Austria (3):
  - Research Site 30043-013, Salzburg
  - Research Site 30043-012, Vienna
  - Research Site 30043-001, Weiz
- Brazil (5):
  - Research Site 30055-036, Curitiba
  - Research Site 30055-021, Porto Alegre
  - Research Site 30055-035, Rio de Janeiro
  - Research Site 30055-025, Salvador
  - Research Site 30055-025, São Paulo
- Chile (10):
  - Research Site 30056-013, Santiago, Providencia
  - Research Site 30056-009, Curicó
  - Research Site 30056-007, Santiago
  - Research Site 30056-013, Santiago
  - Research Site 30056-011, Santiago
  - Research Site 30056-010, Santiago
  - Research Site 30056-006, Santiago
  - Research Site 30056-012, Santiago
  - Research Site 30056-005, Temuco
  - Research Site 30056-014, Viña del Mar
- Research Site 30086-021, Shanghai, China
- Croatia (3):
  - Research Site 30385-008, Zadar
  - Research Site 30385-002, Zagreb
  - Research Site 30385-007, Zagreb
- Czechia (7):
  - Research Site 30420-018, Brno
  - Research Site 30420-012, Brno
  - Research Site 30420-003, Jindřichův Hradec
  - Research Site 30420-007, Lovosice
  - Research Site 30420-014, Olomouc
  - Research Site 30420-010, Strakonice
  - Research Site 30420-009, Teplice
- France (12):
  - Research Site 30033-012, Cholet
  - Research Site 30033-005, Grenoble
  - Research Site 30033-013, Libourne
  - Research Site 30033-014, Lille
  - Research Site 30033-002, Lyon
  - Research Site 30033-001, Marseille
  - Research Site 30033-006, Marseille
  - Research Site 30033-007, Montpellier
  - Research Site 30033-003, Paris
  - Research Site 30033-015, Reims
  - Research Site 30033-004, Saint-Herblain
  - Research Site 30033-018, Strasbourg
- Germany (16):
  - Research Site 30049-081, Augsburg
  - Research Site 30049-060, Berlin
  - Research Site 30049-005, Berlin
  - Research Site 30049-004, Cottbus
  - Research Site 30049-082, Delitzsch
  - Research Site 30049-059, Frankfurt
  - Research Site 30049-019, Frankfurt
  - Research Site 30049-006, Fürstenwalde
  - Research Site 30049-035, Hanover
  - Research Site 30049-073, Homburg
  - Research Site 30049-061, Leipzig
  - Research Site 30049-056, Leipzig
  - Research Site 30049-038, Magdeburg
  - Research Site 30049-051, Munich
  - Research Site 30049-028, Munich
  - Research Site 30049-029, Witten
- Hungary (7):
  - Research Site 30036-005, Balassagyarmat
  - Research Site 30036-001, Budapest
  - Research Site 30036-014, Debrecen
  - Research Site 30036-017, Edelény
  - Research Site 30036-013, Gödöllő
  - Research Site 30036-006, Szeged
  - Research Site 30036-018, Szigetvár
- India (11):
  - Research Site 30091-006, Ahmedabad, Gujarat
  - Research Site 30091-010, Ahmedabad, Gujarat
  - Research Site 30091-011, Himmatnagar, Gujarat
  - Research Site 30091-001, Surat, Gujarat
  - Research Site 30091-024, Rohtak, Haryana
  - Research Site 30091-043, Aurangabad, Maharashta
  - Research Site 30091-004, Nagpur, Maharashta
  - Research Site 30091-023, Nagpur, Maharashta
  - Research Site 30091-033, Pune, Maharashta
  - Research Site 30091-018, Jaipur, Rajasthan
  - Research Site 30091-021, Kanpur
- Israel (6):
  - Research Site 30972-008, Beersheba
  - Research Site 30972-001, Jerusalem
  - Research Site 30972-009, Kfar Saba
  - Research Site 30972-011, Ramat Gan
  - Research Site 30972-012, Rehovot
  - Research Site 30972-005, Sha‘ar Ha‘Aliya
- Italy (7):
  - Research Site 30039-004, Bergamo
  - Research Site 30039-012, Ferrara
  - Research Site 30039-020, Genova
  - Research Site 30039-013, Napoli
  - Research Site 30039-002, Padua
  - Research Site 30039-017, Reggio Emilia
  - Research Site 30039-011, Roma
- Research Site 20081-010, Kanazawa, Japan
- Lithuania (3):
  - Research Site 30370-016, Kaunas
  - Research Site 30370-017, Klaipėda
  - Research Site 30370-002, Vilnius
- Mexico (7):
  - Research Site 30052-024, Guadalajara, Jalisco
  - Research Site 30052-025, Morelia, Michoacon
  - Research Site 30052-026, Chihuahua City
  - Research Site 30052-030, Durango
  - Research Site 30052-033, León
  - Research Site 30052-028, Mexico City
  - Research Site 30052-023, Monterrey
- Peru (7):
  - Research Site -30051-023, Arequipa
  - Research Site 30051-022, Lima
  - Research Site 30051-026, Lima
  - Research Site 30051-020, Lima
  - Research Site -30051-028, Lima
  - Research Site 30051-017, Lima
  - Research Site 30051-021, Lima
- Puerto Rico (4):
  - Research Site 30787-388, Rio Piedras
  - Research Site 30001-383, San Juan
  - Research Site 30787-405, San Juan
  - Research Site 30001-345, Vega Baja
- South Africa (21):
  - Research Site 30027-013, Benoni
  - Research Site 30027-009, Cape Town
  - Research Site 30027-011, Cape Town
  - Research Site 30027-012, Cape Town
  - Research Site 30027-021, Cape Town
  - Research Site 30027-007, Durban
  - Research Site 30027-001, Durban
  - Research Site 30027-014, Durban
  - Research Site 30027-023, Durban
  - Research Site 30027-010, Durban
  - Research Site 30027-030, Johannesburg
  - Research Site 30027-026, Johannesburg
  - Research Site 30027-031, Krugersdorp
  - Research Site 30027-008, KwaZulu
  - Research Site 30027-032, Plettenberg Bay
  - Research Site 30027-029, Polokwane
  - Research Site 30027-004, Pretoria
  - Research Site 30027-019, Pretoria
  - Research Site 30027-015, Thabazimbi
  - Research Site 30027-018, Vereeniging
  - Research Site 30027-017, Welkom
- South Korea (6):
  - Research Site 30082-019, Gwangju
  - Research Site 30082-022, Seoul
  - Research Site 30082-018, Seoul
  - Research Site 20082-028, Seoul
  - Research Site 30082-010, Suwon
  - Research Site 30082-017, Wŏnju
- Spain (12):
  - Research Site 30034-046, A Coruña
  - Research Site 30034-052, A Coruña
  - Research Site 30034-011, Barcelona
  - Research Site 30034-049, Barcelona
  - Research Site 30034-013, Barcelona
  - Research Site 30034-021, Lugo
  - Research Site 30034-053, Madrid
  - Research Site 30034-037, Madrid
  - Research Site 30034-045, Madrid
  - Research Site 30034-050, Santander
  - Research Site 30034-043, Valencia
  - Research Site 30034-041, Vigo
- Taiwan (10):
  - Research Site 30886-013, Douliu
  - Research Site 30886-004, New Taipei City
  - Research Site 30886-006, New Taipei City
  - Research Site 30886-005, Taichung
  - Research Site 30886-007, Taichung
  - Research Site 30886-011, Tainan
  - Research Site 30886-010, Taipei
  - Research Site 30886-008, Taipei
  - Research Site 30886-003, Taipei
  - Research Site 30886-009, Taipei
- Turkey (Türkiye) (18):
  - Research Site 30090-017, Alanya
  - Research Site 30090-018, Ankara
  - Research Site 30090-021, Ankara
  - Research Site 30090-008, Ankara
  - Research Site 30090-009, Ankara
  - Research Site 30090-029, Antalya
  - Research Site 30090-019, Bornova
  - Research Site 30090-016, Çanakkale
  - Research Site 30090-027, Gaziantep
  - Research Site 30030-024, Istanbul
  - Research Site 30090-020, Istanbul
  - Research Site 30090-026, Istanbul
  - Research Site 30090-011, Istanbul
  - Research Site 30090-012, Izmir
  - Research Site 30090-013, Mersin
  - Research Site 30090-010, Nilufer
  - Research Site 30090-022, Tekirdağ
  - Research Site 30090-002, Yüreğir
- Ukraine (2):
  - Research Site 30380-002, Chernivtsi
  - Research Site 30380-011, Kyiv
- United Kingdom (4):
  - Research Site 30044-027, Glasgow
  - Research Site 30044-059, High Wycombe
  - Research Site 30044-039, Leicester
  - Research Site 30044-025, Sheffield

IPD SHARING:
Plan to Share IPD: No